CLINICAL TRIAL: NCT06386315
Title: Reduced Dose Hypofractionated Radiotherapy (3Gy x 3 Fractions) for Indolent Non-Hodgkin Lymphoma (POSEIDON): A Multisite Phase 2 Randomized Trial
Brief Title: Reduced Dose Radiotherapy for the Treatment of Indolent Non-Hodgkin Lymphoma
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Mayo Clinic (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MC230808; NCI-2024-03242 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 23-010273 (Other: Mayo Clinic Institutional Review Board); MC230808 (Other: Mayo Clinic)
Record Dates: First submitted 2024-04-23; First posted 2024-04-26 (Actual); Last update posted 2025-11-24 (Actual); Status verified 2025-11

CONDITIONS: Indolent B-Cell Non-Hodgkin Lymphoma; Recurrent Indolent B-Cell Non-Hodgkin Lymphoma; Refractory Indolent B-Cell Non-Hodgkin Lymphoma; Recurrent Indolent Non-Hodgkin Lymphoma; Refractory Indolent Non-Hodgkin Lymphoma
MeSH Terms: interventions — Endoscopy; Magnetic Resonance Spectroscopy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- ARM 1 (reduced dose ISRT) (Experimental): Patients undergo reduced dose ISRT once daily (excluding weekends): 9 Gy delivered in 3 treatment fractions or 8 Gy in 2 fractions. At physician discretion, patients may receive 10 Gy in 5 fractions. Patients also undergo CT or PET/CT throughout the study. Patients may additionally undergo endoscopy during screening and during follow up.
  Interventions: Procedure: Computed Tomography; Procedure: Endoscopic Procedure; Radiation: Involved-site Radiation Therapy (3 Fractions); Procedure: Positron Emission Tomography; Other: Questionnaire Administration
- ARM 2 (SOC ISRT) (Active Comparator): Patients undergo standard of care (SOC) radiation therapy once daily (excluding weekends): 24 Gy in 12 treatment fractions. Patients also undergo CT or PET/CT throughout the study. Patients may additionally undergo endoscopy during screening and during follow up.
  Interventions: Procedure: Computed Tomography; Procedure: Endoscopic Procedure; Radiation: Involved-site Radiation Therapy (12 Fractions); Procedure: Positron Emission Tomography; Other: Questionnaire Administration

INTERVENTIONS:
Procedure: Computed Tomography — Undergo CT or PET/CT
  Other Names: CAT; CAT Scan; Computed Axial Tomography; Computerized Axial Tomography; Computerized axial tomography (procedure); Computerized Tomography; Computerized Tomography (CT) scan; CT; CT Scan; tomography
Procedure: Endoscopic Procedure — Undergo endoscopy
  Other Names: Endoscopic Examination; Endoscopy; ES
Radiation: Involved-site Radiation Therapy (3 Fractions) — Undergo ISRT in 3 fractions
  Other Names: ISRT
  Arms: ARM 1 (reduced dose ISRT)
Radiation: Involved-site Radiation Therapy (12 Fractions) — Undergo ISRT in 12 fractions
  Other Names: ISRT
  Arms: ARM 2 (SOC ISRT)
Procedure: Positron Emission Tomography — Undergo PET/CT
  Other Names: Medical Imaging, Positron Emission Tomography; PET; PET Scan; Positron emission tomography (procedure); Positron Emission Tomography Scan; Positron-Emission Tomography; proton magnetic resonance spectroscopic imaging; PT
Other: Questionnaire Administration — Ancillary studies

SUMMARY:
This phase II trial compares the safety, side effects and effectiveness of reduced dose radiation therapy to standard of care dose radiation in treating patients with indolent non-Hodgkin lymphoma. Radiation therapy uses high energy x-rays, particles, or radioactive seeds to kill cancer cells and shrink tumors. Standard of care radiation treatment for indolent non-Hodgkin lymphoma is usually delivered in 12 treatments. Studies have shown indolent lymphoma to be sensitive to radiation treatment, however, larger doses have higher rates of toxicities. A reduced radiation dose may be safe, tolerable and/or effective compared to standard of care radiation dose in treating patients with indolent non-Hodgkin lymphoma.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To show that the experimental arm [9 gray (Gy) in 3 fractions, 8 Gy in 2 fractions, or 10 Gy in 5 fractions] has significantly reduced acute toxicity (grade ≥ 2 adverse events at least possibly related to radiation treatment within 14 days after the end of radiation treatment [according to Common Terminology Criteria for Adverse Events (CTCAE) version (v)5.0] compared to 24 Gy in 12 fractions.

SECONDARY OBJECTIVES:

I. To evaluate patient reported quality of life. II. To evaluate response rate. III. To evaluate local control rate. IV. To evaluate relapse-free survival.

EXPLORATORY OBJECTIVES:

I. Financial toxicity will be assessed at the end of radiation treatment. II. Financial health care expenditure will be assessed at the end of radiation treatment III. Late toxicity.

CORRELATIVE RESEARCH OBJECTIVES:

I. Biopsies of enrolled patients will be evaluated for pathological assessment of cellular and genetic mutations to correlate them with disease local relapse and radiation resistance.

II. Patients will have their baseline positron emission tomography (PET)/computed tomography (CT) scan undergo auto-segmentation to calculate the functional imaging 18-fluoro-deoxyglucose (FDG) metabolic tumor volume (MTV), total lesions glycolysis (TLG) and maximum standardized uptake volume (SUVmax) of the sites to be treated with involved-site radiation therapy (ISRT) using MIMvista platform to correlate it with disease local relapse and treatment response.

OUTLINE: Patients are randomized to 1 of 2 arms.

ARM I: Patients undergo reduced dose ISRT once daily (QD) over 3, 2, or 5 treatment fractions. Patients also undergo CT or PET/CT throughout the study. Patients may additionally undergo endoscopy during screening and during follow up.

ARM II: Patients undergo standard of care (SOC) radiation therapy QD over 12 treatment fractions. Patients also undergo CT or PET/CT throughout the study. Patients may additionally undergo endoscopy during screening and during follow up.

After completion of study treatment, patients are followed up at days 7 and 14, months 3 and 6, and then every 6 months for up to 2 years post-radiation therapy.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* Histological confirmation of indolent B-cell lymphoma that can include any of the following:

  * Follicular lymphoma (grade 1 or 2 or 3A)
  * Marginal zone lymphoma (nodal or extranodal)
  * Follicle center lymphoma
* Any stage disease
* Initial, refractory, or relapsed disease. If relapse involves the site to be treated there must be evidence of disease progression
* Eastern Cooperative Oncology Group (ECOG) performance status (PS) ≤ 3
* Negative pregnancy test done ≤ 7 days prior to registration, for persons of childbearing potential only
* Provide written informed consent
* Ability to complete questionnaire(s) by themselves or with assistance
* Willing to return to enrolling institution for follow-up visits (during the active monitoring phase of the study). Virtual visits can also be considered as an option for applicable items
* Confirmation from radiation oncologist of suitability to participate in study

Exclusion Criteria:

* Any of the following:

  * Pregnant women
  * Nursing women
  * Women of childbearing potential who are unwilling to employ adequate contraception
* T-cell lymphoma
* Receiving treatment for small and chronic lymphocytic lymphoma
* Grade 3B follicular lymphoma

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 112 (Estimated)
Dates: Start 2024-05-15 (Actual); Primary Completion 2026-05-30 (Estimated); Study Completion 2026-05-30 (Estimated)

PRIMARY OUTCOMES:
Incidence of grade 2 or higher acute adverse events (AEs) | Up to 14 days after radiation treatment
  AEs will be graded using Common Terminology Criteria for Adverse Events (CTCAE) version 5.0. Acute toxicity will be reported as a proportion calculated as the number of patients with acute toxicity divided by the total number of treatment patients. Treatment cycles are 5 days ±2 days (Arm 1) and 16 days ±2 days (Arm 2).

SECONDARY OUTCOMES:
Response rate | Up to 3 months after radiation treatment
  Response rate will be defined as the proportion of patients displaying response (complete response or partial response) at 3 months post treatment. Complete response is defined as the disappearance of all signs of cancer in response to treatment. Partial response is defined decrease in the size of target lesions by ≥ 50%, with no increase in the size of any lesion and no appearance of new lesions. Treated patients who do not have a 3-month evaluation will be classified as a non-response. Treatment cycles are 5 days ±2 days (Arm 1) and 16 days ±2 days (Arm 2).
Time to progression rate | Up to 24 months after radiation treatment
  Local control will be defined as the number of days from end of radiation treatment until first local recurrence within 24 months post radiation treatment. Treatment cycles are 5 days ±2 days (Arm 1) and 16 days ±2 days (Arm 2).
Patient reported quality of life | Up to 3 months after radiation treatment
  Patient reported quality of life will be measured using Functional Assessment of Chronic Illness Therapy-Fatigue (FACIT-F) scale, a 13-item questionnaire answered on a scale of 1-5 where 1=Not at all and 5=Very much. Treatment cycles are 5 days ±2 days (Arm 1) and 16 days ±2 days (Arm 2).

CONTACTS AND LOCATIONS:
Overall Officials: Bradford S. Hoppe, MD, MPH, Principal Investigator — Mayo Clinic
Locations (7):
- United States (7):
  - Mayo Clinic in Arizona, Scottsdale, Arizona
  - Mayo Clinic in Florida, Jacksonville, Florida
  - Mayo Clinic Health System in Albert Lea, Albert Lea, Minnesota
  - Mayo Clinic Health System - Mankato, Mankato, Minnesota
  - Mayo Clinic in Rochester, Rochester, Minnesota
  - Mayo Clinic Health System-Eau Claire Clinic, Eau Claire, Wisconsin
  - Mayo Clinic Health System-Franciscan Healthcare, La Crosse, Wisconsin

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials